CLINICAL TRIAL: NCT00808743
Title: Prevention of Progression of Duodenal Adenomas to Cancer in Patients With Familial Adenomatous Polyposis (FAP)
Brief Title: Prevention of Progression of Duodenal Adenomas in Patients With Familial Adenomatous Polyposis
Acronym: PreDuoFAP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RUN 2008-4198; ABR nr.: NL23569.091.08; CMO: 2008/148; EudraCT: 2008-003696-43
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2010-08

CONDITIONS: Familial Adenomatous Polyposis; Duodenal Neoplasms; Duodenal Polyps
Keywords: Familial adenomatous polyposis; Adenomatous Polyposis Coli; Digestive System Neoplasms; Gastrointestinal Disease; Intestinal disease; Intestinal neoplasms; Gastrointestinal neoplasms; Polyps; Adenoma; Adenomatous Polyps; Neoplastic Syndromes, Hereditary; Digestive System Diseases; Genetic Diseases, Inborn; Chemoprevention; Celecoxib; Ursodeoxycholic acid; Anti-Inflammatory agents, Non-Steroidal; Cyclooxygenase Inhibitors
MeSH Terms: conditions — Adenomatous Polyposis Coli; Duodenal Neoplasms; Digestive System Neoplasms; Gastrointestinal Diseases; Intestinal Diseases; Intestinal Neoplasms; Gastrointestinal Neoplasms; Polyps; Adenoma; Adenomatous Polyps; Neoplastic Syndromes, Hereditary; Digestive System Diseases; Genetic Diseases, Inborn | interventions — Celecoxib; Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Patients receive oral celecoxib twice daily and oral placebo twice daily
  Interventions: Drug: Celecoxib; Drug: Placebo
- Group 2 (Experimental): Patients receive oral celecoxib twice daily and oral ursodeoxycholic acid twice daily
  Interventions: Drug: Celecoxib; Drug: Ursodeoxycholic acid

INTERVENTIONS:
Drug: Celecoxib — Celecoxib: 400mg twice daily, orally, 6 months
Drug: Ursodeoxycholic acid — Ursodeoxycholic acid: orally, 6 months, dosage based on body weight:
  below 50 kg: 1000mg, divided in two daily doses; 50-70 kg: 1500mg, divided in two daily doses; over 70 kg: 2000mg, divided in two daily doses
  Arms: Group 2
Drug: Placebo — Placebo: orally, 6 months, dosage based on body weight:
  below 50 kg: 1000mg, divided in two daily doses; 50-70 kg: 1500mg, divided in two daily doses; over 70 kg: 2000mg, divided in two daily doses
  Arms: Group 1

SUMMARY:
Duodenal carcinomas are the leading cause of mortality in patients with Familial Adenomatous Polyposis (FAP) who underwent prophylactic colorectal surgery. The purpose of this study is to determine wether celecoxib combined with ursodeoxycholic acid is an effective chemoprevention strategy to influence the progression of duodenal adenomas to carcinomas in patients with FAP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Familial adenomatous Polyposis: APC-mutation identified or more than 100 colorectal polyps on diagnosis
* Spigelman score of duodenal adenoma equal to II or III

Exclusion Criteria:

* Incapability of signing informed consent
* Active gastric or duodenal ulcer, gastrointestinal bleeding
* Cardiovascular disease or risk:

  * Congestive cardiac failure: NYHA class II to IV
  * Proven ischemic heart disease and/or cerebrovascular disease
  * Risk factors: hypertension, hyperlipidaemia, diabetes mellitus, family history of cardiovascular events (≥2 first degree family members <55 years)
* Renal dysfunction: creatinine clearance below 50mL/min
* Liver dysfunction: albumin below 25 g/L or Child-Pugh-score equal to or below 10
* Known allergic reaction to sulfonamides, NSAIDs or ursodeoxycholic acid
* Use of NSAIDs or ursodeoxycholic acid for more than 1 week during the 6 months prior to the start of the study
* Use of lithium
* Symptomatic gallstones
* Inflammatory bowel disease
* (Possible) pregnancy or breast feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-05; Primary Completion 2011-07 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in number and size of duodenal adenomas (assessed directly and by evaluation of video and photographic material from endoscopic procedures) | Baseline, 6 months

SECONDARY OUTCOMES:
Cell proliferation, in normal mucosa and adenomas (if present) | Baseline, 6 months
Biliary acid profile (if present) | Baseline, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Fokko M Nagengast, MD, Ph D, Principal Investigator — University Medical Center St. Radboud Nijmegen, The Netherlands; Bjorn WH van Heumen, MD, Principal Investigator — University Medical Center St. Radboud Nijmegen, The Netherlands; Wilbert HM Peters, Ph D, Principal Investigator — University Medical Center St Radboud Nijmegen, The Netherlands; Ellen Kampman, Ph D, Principal Investigator — University Medical Center St Radboud Nijmegen, The Netherlands
Locations (5):
- Netherlands (5):
  - Academic Medical Center, Amsterdam
  - University Medical Center, Groningen
  - Leiden University Medical Center, Leiden
  - University Medical Center St. Radboud, Nijmegen
  - Erasmus Medical Center, Rotterdam

REFERENCES:
- [Derived] van Heumen BW, Roelofs HM, te Morsche RH, Nagengast FM, Peters WH. Duodenal mucosal risk markers in patients with familial adenomatous polyposis: effects of celecoxib/ursodeoxycholic acid co-treatment and comparison with patient controls. Orphanet J Rare Dis. 2013 Nov 19;8:181. doi: 10.1186/1750-1172-8-181. PMID 24245549
- [Derived] van Heumen BW, Roelofs HM, Vink-Borger ME, Dekker E, Mathus-Vliegen EM, Dees J, Koornstra JJ, Langers AM, Nagtegaal ID, Kampman E, Peters WH, Nagengast FM. Ursodeoxycholic acid counteracts celecoxib in reduction of duodenal polyps in patients with familial adenomatous polyposis: a multicentre, randomized controlled trial. Orphanet J Rare Dis. 2013 Aug 6;8:118. doi: 10.1186/1750-1172-8-118. PMID 23919274